CLINICAL TRIAL: NCT00015483
Title: Hematotoxic Effects of Benzene and Doxorubicin
Brief Title: Hematotoxic Effects of Particulate Exposure
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 5020-CP-001
Record Dates: First submitted 2001-04-20; First posted 2001-04-23 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Cancer
Keywords: Hematotoxicity; Benzene; Bone Marrow
MeSH Terms: conditions — Neoplasms

SUMMARY:
Hematotoxicity is caused by a number of agents such as a benzene by-product called hydroquinone and the antitumor agent doxorubicin. This is a basic research study, conducted using normal human donors, of mechanisms involved in hematotoxicity and of the protective response of human hematopoietic progenitor cells to hematotoxic agents. Tumor necrosis factor exposure protects these cells from a subsequent exposure to hematotoxic agents. The alteration of gene expression in these cells caused by tumor necrosis factor is being studied. Additionally, the tumor necrosis factor-induced biochemical pathways involved in protection of human hematopoietic progenitor cells will be studied.

ELIGIBILITY:
* healthy
* nonsmoking
* no history of hematologic disorder
* not pregnant
* no medications which suppress hematopoiesis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult